CLINICAL TRIAL: NCT05270343
Title: The Effect of Early High-dose Vitamin D Intervention on the Residual β-cell Function in Adolescents and Children With Type 1 Diabetes
Brief Title: Early High-Dose Vitamin D and Residual β-Cell Function in Pediatric Type 1 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Weiqiong Gu, The Effect of Early High-dose Vitamin D Intervention on the Residual β-cell Function in Adolescents and Children With Type 1 Diabetes, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YZhang
Record Dates: First submitted 2022-02-25; First posted 2022-03-08 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Experimental): In 99 subjects of 3-18yr with newly-onset T1D, oral administration of 140IU/kg qd of cholecalciferol will be given until the serum 25(OH)D3 was maintained at the upper limit of normal range(50-80 ng/ml[125-200 nmol/L], ≤100 ng/ml[≤250 nmol/L]) for the loading peroid. And then oral administration of 70IU/kg qd of cholecalciferol for the maintenance period, meanwhile combined with intensive Insulin therapy for 12 months.
  Interventions: Drug: Cholecalciferol (Vit D3) 400Unit Cap
- Insulin (No Intervention): In 99 subjects of 3-18yr with newly-onset T1D, only intensive insulin therapy will be given for 12 months.

INTERVENTIONS:
Drug: Cholecalciferol (Vit D3) 400Unit Cap — Each subject will take Vit D3 (400Unit Cap) with breakfast for 12 consecutive months, and the initial load will be 140IU/kg qd until the serum 25(OH)D3 is maintained at the upper limit of normal ( 50-80ng/ml[125-200nmol/L], ≤100ng/ml[≤250nmol/L]), then maintained at 70IU/kg qd, combined with intensive insulin therapy
  Other Names: Cholecalciferol
  Arms: Vitamin D

SUMMARY:
The project aims to study the effect of early high-dose vitamin D supplementation on type 1 diabetes in children and adolescents receiving intensive insulin therapy. The results may lead to major changes in the early treatment of type 1 diabetes, with special emphasis on the use of vitamin D to improve the function of residual β-cells and maintain standardized insulin therapy for these patients. The overall goal is to reduce the long-term complications of type 1 diabetes.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is a chronic autoimmune disease that is immune-mediated destruction of pancreatic β-cells. It relies on insulin therapy. The currently accepted standardized treatment is intensive insulin therapy (>3 injections per day). The incidence of T1D is increasing globally, prompting researchers to study new immune regulation strategies to stop the autoimmune process and change the progression of the disease. T1D is considered to be a multifactorial disease, where genetic susceptibility and environmental factors interact to promote the triggering of an autoimmune response against β cells. In the past few decades, in addition to the established role of vitamin D in regulating calcium homeostasis and bone metabolism, vitamin D also played an anti-inflammatory and immunomodulatory role in inflammation. In addition, the global incidence of vitamin D deficiency is also increasing sharply, providing epidemiological evidence for the involvement of T1D vitamin D deficiency in the pathogenesis. Polymorphisms in key genes involved in vitamin D metabolism have also been shown to regulate the risk of T1D.

The results of animal experiments show that vitamin D can preserve the number and function of β cells through different mechanisms, such as: (1) promoting the transition from Th1 to Th2 cytokine expression profile, (2) enhancing the clearance of autoreactive T cells and reducing pancreatic islets infiltration of Th1 cells, (3) reducing cytokine-induced β cell damage, and the major histocompatibility complex (MHC) class I and II expression in β cells, (4) promoting Tregs differentiation and inhibition ability. Different intervention studies and randomized controlled trials have shown that supplementation of cholecalciferol (vitamin D3-a safe and easy-to-implement treatment for children, with a toxic dose of 20,000 to 50,000 IU/d for infants and young children and continuously taken for several weeks) in T1D patients can protect residual β Cell function (RBCF) and improve glycemic control: Gabbay et al. found that patients with newly-onset T1D receiving oral vitamin D3 (2000 IU/day) for 18 months can effectively slow down the rate of decrease in C-peptide levels after meals. In addition, the level of glycated hemoglobin (HbA1c) decreases; vitamin D3 (3000 IU/day) treatment for 12 months can delay the decline of RBCF in children with T1D within 1-2 years of the disease course and improve glycemic control. However, some reports found that according to age groups (1-3 years old -60,000 IU, 4-8 years old -90,000 IU, 9-18 years old-1,20,000 IU), with oral vitamin D3 administered once a month for 6 consecutive months, although it can improve fasting C-peptide (FCP) levels, it did not reduce HbA1c and daily insulin requirements; Perchard et al. proved that a single oral vitamin D3 (100,000 or 160,000 IU) failed to improve HbA1c levels in children with T1D.

Based on the results of previous studies, some researchers believe that maintaining a stable serum 25(OH)D3 level at an adequate level of vitamin D (>30/mL[>75 nmol/L]) may be more meaningful than a single high-dose oral vitamin D3. The latter is likely to be unable to maintain sufficient serum 25(OH)D3 levels during long-term follow-up. Therefore, Treiber et al. gave 15 children with newly-onset T1D oral vitamin D3 (70 IU/kg/d-first month loading dose 140 IU/kg/d) for 12 consecutive months to maintain a high level of serum 25(OH)D3. Compared with the placebo group, the intervention group had better peripheral blood Treg function at 12 months, but there was no significant difference in islet function and HbA1c level between the two groups (in intervention group, the percentage of 25(OH)D3 level>50 ng/mL[> 125 nmol/L]) was 50% after 3 months while 36% after 12 months); some researchers use direct supplementation of 25(OH)D3 (calcifediol), starting at 10ug/d until the serum 25(OH)D3 50-80 ng/mL[125-200 nmol/L] level is maintained (maintained at 71±5 ng/mL[177.5±12.5 nmol/L] after 1 year on average), FCP level of the intervention group remained stable after 1 year of treatment ; some studies have used calcitriol (1,25(OH)D3, or active vitamin D) 0.25ug qod for continuous oral administration for 1 year. The insulin consumption of the intervention group decreased, but no difference was observed in islet function.

It's worth noting that an individual's response to a given dose of vitamin D is highly variable and depends on several factors, such as baseline vitamin D status, body fat percentage, gender, ethnicity, genetics, seasonal changes, medications, and vitamin D formula type. Therefore, the optimized research design is necessary to more effectively evaluate the impact of vitamin D on the research results. Cholecalciferol (vitamin D3) is still considered the most promising vitamin D dosage form due to its long half-life, large safety window, and convenience (over-the-counter medication). To sum up, this study intends to use cholecalciferol, integrated individual factors, on the basis of maintaining a high serum 25(OH)D3 level, and an optimized research plan to extend the intervention time to evaluate the effect of vitamin D on T1D pancreatic islet function.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 3-18 years
2. Sex: male and female participants will be enrolled
3. Immune-mediated T1D: presence of at least one diabetes-associated autoantibody (ADA 2021 guideline for reference)
4. T1D duration of <6 months (from first diagnosis of T1D)
5. Fasting C-peptide level (FCP) of >0.1 nmol/L (0.3ng/mL) ; or 2-hour post-meal stimulated C-peptide level (PCP) of ≥ 0.2 nmol/L(0.6 ng/mL)(with mixed meal tolerance test, MMTT)
6. Vitamin D deficiency: baseline 25(OH)D3< 30 ng/mL (<75 nmol/L)

Exclusion Criteria:

1. Participants with severe chronic and systemic diseases: tumors, immunodeficiency, arteriosclerosis, heart failure, hypercholesterolemia, kidney disease
2. Participants with calcium and phosphorus metabolism disorders
3. Participants on medications or dietary supplements that affect Ca or Vitamin D in the past 6 months
4. Participants on medications other than insulin that can affect blood glucose level
5. Participants with malabsorption
6. Participants with infectious diseases
7. Participants with mental illness
8. The receipt of any investigational drug within 6 months prior to this trial

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 198 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Residual β-Cell function (RBCF) | 12 months
  To study the effect of early supplementation of high-dose vitamin D on RBCF in the first 12 months after diagnosis of T1D by using fasting C-peptide(FCP) levels to quantify RBCF across longitudinal measurements

SECONDARY OUTCOMES:
Glycemic control (HbA1c) | 12 months
  To study the effect of early supplementation of high-dose vitamin D on glycemic control by comparing HbA1c values across longitudinal measurements
Glycemic control (free blood glucose) | 12 months
  To study the effect of early supplementation of high-dose vitamin D on glycemic control by comparing free blood glucose (FBG) values across longitudinal measurements
Glycemic control (postprandial blood glucose) | 12 months
  To study the effect of early supplementation of high-dose vitamin D on glycemic control by comparing postprandial blood glucose (PBG) values across longitudinal measurements
Islet Function (stimulated C-peptide) | 12 months
  To study the effect of early supplementation of high-dose vitamin D on the reserve capacity of RBCF by using 2-hour post-meal stimulated C peptide (PCP) with mixed meal tolerance test (MMTT) across longitudinal measurements
Daily Insulin Dosage | 12 months
  To study the effect of early supplementation of high-dose vitamin D on the insulin requirement by using daily insulin dosage per body weight (DID IU/kg.d) across longitudinal measurements

CONTACTS AND LOCATIONS:
Overall Officials: Zhiya Dong, Principal Investigator — Department of Pediatrics, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Department of Pediatrics, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China